CLINICAL TRIAL: NCT05597059
Title: The Diagnostic Value of the First Clinical Impression of Patients Presenting to the Emergency Department
Brief Title: The Diagnostic Value of the First Clinical Impression of Patients Presenting to the Emergency Department (PREKEYDIA)
Status: Completed | Type: Observational
Sponsor: Kepler University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PREKEYDIA
Record Dates: First submitted 2022-10-25; First posted 2022-10-27 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Shortness of breath
  Interventions: Diagnostic Test: Machine Learning Prediction
- Extremity pathologies
  Interventions: Diagnostic Test: Machine Learning Prediction
- Abdominal pain
  Interventions: Diagnostic Test: Machine Learning Prediction
- Urological pathologies
  Interventions: Diagnostic Test: Machine Learning Prediction
- Chest pain
  Interventions: Diagnostic Test: Machine Learning Prediction
- Back pain
  Interventions: Diagnostic Test: Machine Learning Prediction

INTERVENTIONS:
Diagnostic Test: Machine Learning Prediction — Machine Learning Prediction

SUMMARY:
Finding a diagnosis for acutely ill patients places high demands on emergency medical personnel. While anamnesis and clinical examination provide initial indications and allow a tentative diagnosis, both laboratory chemistry and imaging tests are used to confirm (or exclude) the tentative diagnosis. The more precise and targeted the additional laboratory chemical or radiological diagnosis, the more quickly and economically the causal treatment of the emergency patient can be initiated.

One examination modality, which in addition to the medical history and clinical examination, could quickly provide information about the condition of the patient, their clinical picture and severity of illness, is the first clinical impression of the patient (so-called "first impression" or "end-of-bed view"). This describes the first sensory impression that the medical staff gathers from a patient. This includes visual (e.g., facial expression, gait, breathing), auditory (e.g., voice pitch, shortness of breath when speaking), and olfactory (e.g., smell of exhaled air, body odor) impressions. Clinical practice shows that a great deal of important additional information can be gathered through this first clinical impression, which, together with the history and clinical examination of the emergency patient, provides valuable clues to the underlying condition.

To date, however, only scattered data and study results exist in the medical literature on the value of the first clinical impression in the care of emergency patients. In the present prospective observational study, the study attempts to evaluate the predictive value of the first clinical impression in identifying a leading symptom and other important clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the emergency department between 2019-09-01 and 2020-02-28.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults presenting to the emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 1506 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
AUROC for Classification of Shortness of Breath | 2019-09-01 to 2020-02-28
  AUROC for Classification of Shortness of Breath
AUROC for Classification of Extremity Pathologies | 2019-09-01 to 2020-02-28
  AUROC for Classification of Extremity Pathologies
AUROC for Classification of Abdominal Pain | 2019-09-01 to 2020-02-28
  AUROC for Classification of Abdominal Pain
AUROC for Classification of Urological Pathologies | 2019-09-01 to 2020-02-28
  AUROC for Classification of Urological Pathologies
AUROC for Classification of Chest Pain | 2019-09-01 to 2020-02-28
  AUROC for Classification of Chest Pain
AUROC for Classification of Back Pain | 2019-09-01 to 2020-02-28
  AUROC for Classification of Back Pain

SECONDARY OUTCOMES:
AUROC for Classification of Hospital Admission | 2019-09-01 to 2020-02-28
  AUROC for Classification of Hospital Admission
Confusion Matrix | 2019-09-01 to 2020-02-28
  Confusion Matrix Results: true positives, true negatives, false positive, false negatives and values calculated from these results.
Descriptive Statistics | 2019-09-01 to 2020-02-28
  Descriptive Statistics (e. g. age in years)

CONTACTS AND LOCATIONS:
Locations (1):
- Kepler University Hospital, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No